CLINICAL TRIAL: NCT06344169
Title: Efficacy of Parenteral Injection of an Extended Release Kappa-receptor Opioid Sebacoyl Dinalbuphine Ester for Pain Management After Cesarean Section: a Randomized, Open-label, Non-inferiority Trial
Brief Title: Dinalbuphine Ester (Naldebain) for Pain Management After Cesarean Section
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTCRD112(2)-I-15
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-02

CONDITIONS: Postsurgical Pain; Cesarean Section; Chronic Post-surgical Pain
Keywords: kappa agonist; mu agonist; Intrathecal morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — sebacoyl dinalbuphine ester; Morphine

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ITM group (Active Comparator): Participants assigned to intrathecal morphine (ITM) group will receive intrathecal injection of morphine (0.15mg) for post-cesarean section pain
  Interventions: Drug: Morphine
- SDE group (Experimental): Participants assigned to sebacoyl dinalbuphine ester (SDE) group will receive intramuscular injection of SDE (150mg) for post-cesarean section pain
  Interventions: Drug: Sebacoyl Dinalbuphine Ester

INTERVENTIONS:
Drug: Sebacoyl Dinalbuphine Ester — SDE will be dissolved in benzyl benzoate and sesame oil (a total volume of 2ml) will be prepared in a 5-ml syringe 30 min before administration. Intramuscular injection into the gluteal muscles will be performed by an anesthesiologist under sonography-guidance
  Other Names: Naldebain
  Arms: SDE group
Drug: Morphine — A single dose of morphine (0.15mg) will be administered along with bupivacaine during spinal anesthesia.
  Arms: ITM group

SUMMARY:
Inadequate postoperative pain management can lead to physical and psychological distress in patients as well as impact surgical wound healing and increase the risk of developing postoperative delirium and cardiopulmonary and thromboembolic events. Severe postoperative pain may also result in the development of chronic post-surgical pain (CPSP), which in turn can lead to prolonged use of opioids and increased health-care costs. A descriptive survey study in 60 postpartum women who received cesarean section suggested that the presence of postoperative pain significantly reduced the willingness of breastfeeding and infant care. The incidence of CPSP after cesarean delivery has been reported to vary from 1% to 18% up to 1 year after operation. Intrathecal morphine (ITM) injection is considered as the standard pain management strategy for post-cesarean pain. However, the overall analgesic effect of ITM is about 8-12h and it is associated with pruritus, nausea/vomiting, urinary retention, constipation, mental status change, and respiratory depression. Therefore, the development of a safe, conveniently operated, and long-lasting analgesic strategy, which serves as background pain control modality up to several days after cesarean section should provide clinically beneficial advantages in the management of acute postoperative pain and prevention of CPSP in postpartum women. Naldebain® is prodrug of nalbuphine, which was approved by the Taiwan FDA in 2017. Naldebain® is rapidly hydrolyzed by tissue of plasma esterase to release nalbuphine. The bioavailability of nalbuphine following intramuscular injection Naldebain® was 85.4%, and it took approximately 6 days for the complete release of Naldebain® into the blood circulation. Therefore, a single parenteral injection of Naldebain® could provide long lasting analgesic effect in several phase II trials. However, Naldebain® has not been tested in the pain control after cesarean section. Therefore, this PI-initiated prospective, randomized, open-label, non-inferiority trial aims to investigate the clinical efficacy of Naldebain® in management of acute postoperative pain in term parturient who receive elective cesarean section to provide analgesic effect that is not inferior to the standard ITM and prevent the development of CPSP.

DETAILED DESCRIPTION:
Inadequate postoperative pain management can lead to physical and psychological distress in patients as well as impact surgical wound healing and increase the risk of developing postoperative delirium and cardiopulmonary and thromboembolic events. Severe postoperative pain may also result in the development of chronic post-surgical pain (CPSP), which in turn can lead to prolonged use of opioids and increased health-care costs. A descriptive survey study in 60 postpartum women who received cesarean section suggested that the presence of postoperative pain significantly reduced the willingness of breastfeeding and infant care. Furthermore, the incidence of CPSP after cesarean delivery has been reported to vary from 1% to 18% up to 1 year after operation. More specifically, an US nationwide survey reported that 79% of mothers who received cesarean section reported experiencing pain at the incision site in the first two months and 18% had persistent pain at least 6 months after operation. Placement of an epidural catheter can be used for epidural anesthesia during cesarean section and continuous epidural infusions of opioids or combined with local anesthetic after cesarean section can result in high-quality analgesia effect for postpartum and postsurgical pain. Intrathecal injection of morphine (ITM) is considered as the standard pain management strategies for post-cesarean pain in Taiwan. However, correct placement of epidural catheter for effective postoperative pain management is more technical demanding, and accidental dural puncture is associated with increased risk of postdural puncture headache. ITM is associated with severe mu-receptor agonist adverse reactions, such as pruritus, nausea/vomiting, urinary retention, constipation, mental status change, and respiratory depression. Therefore, the development of a safe, conveniently operated, and long-lasting non-mu agonism analgesic strategy, which serves as background pain control modality up to several days after cesarean section should provide clinically beneficial advantages in the management of acute postoperative pain and prevention of development of CPSP in postpartum women.

Sebacoyl dinalbuphine ester Naldebain® (SDE) is prodrug of nalbuphine, which was approved by the Taiwan FDA in 2017. SDE is rapidly hydrolyzed by tissue of plasma esterase to release nalbuphine. The bioavailability of nalbuphine following intramuscular injection SDE was 85.4% with a mean absorption time up to 145 h, and it took approximately 6 days for the complete release of SDE into the blood circulation. Therefore, a single parenteral injection of SDE could provide long lasting analgesic effect in several phase II trials. However, SDE has not been tested in the pain control after cesarean section. Therefore, this PI-initiated prospective, randomized, open-label, non-inferiority trial aims to investigate the clinical efficacy of SDE in management of acute postoperative pain in term parturient who receive elective cesarean section to provide analgesic effect that is not inferior to the standard ITM. A single intramuscular injection of SDE may also prevent the development of CPSP after cesarean delivery, as SDE can provide prolonged analgesic effect for up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* term primipara or multipara who are scheduled for elective cesarean section

Exclusion Criteria:

1. Severe pregnancy-induced complication (such as preeclampsia, eclampsia, poorly control pregnancy-induced hypertension and/or diabetes)
2. High risk for postpartum hemorrhage
3. Contraindicated for neuraxial block
4. Preterm (gestational age< 36 week) delivery
5. Emergency cesarean section
6. After-office hour schedule
7. History of substance abuse
8. Known allergy to nalbuphine, benzyl benzoate or sesame oil
9. Eligible parturient who are not willing to follow the assignment of treatment after randomization

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female puerpera
Enrollment: 120 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Intensity of surgical pain after operation as assessed by visual analogue scale | 5 days after cesarean section
  Visual analogue scale (VAS 1-10, a continuum scale in which 0 represents "no pain" and and 10 represents "worst pain.")
Rescue doses of analgesics administered after operation | 5 days after cesarean section
  Total doses of parenteral administered opioids, NSAIDs, cyclooxygenase-2 inhibitors

SECONDARY OUTCOMES:
Incidence of chronic post-surgical pain | 3 months after cesarean section
  Pain that newly develops after operation and lasts >2 months and other causes of pain are excluded
Satisfaction of living after surgery as assessed by the HRQoL short-form (SF)-12 | 3 months after cesarean section
  Quality of life will be assessed by the HRQoL short-form (SF) Questionnaire, which consists a physical component summary (PCS) and a mental component summary (MCS). The rating scales range from yes-no to likert scales, and the final score of PCS and MCS will be calculated by an algorithm (QualityMetric's SF-12v1®). Scores range from 0 to 100, in which lower scores mean lower health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: NING-SHENG LAI, Study Chair — Buddhist Tzu Chi Hospital
Locations (1):
- Dalin Tzu Chi Hospital, Dalin, Chai-Yi, Taiwan

IPD SHARING:
Plan to Share IPD: No